CLINICAL TRIAL: NCT03947957
Title: Microbial Biomarkers of EArly Pseudomonas Aeruginosa Colonization in CHildren With Cystic Fibrosis
Acronym: BEACH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BEACH (29BRC19.0065)
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Defecation; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Infants will be included between the 2nd visit to the CRCM (about 2 months of age) and the 6th month then they will be followed until the age of 36 months. The pace of visits will be based on the usual follow-up rate of CF infants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- collection of expectoration, stools and blood (Other)
  Interventions: Diagnostic Test: collection of expectoration, stools and blood

INTERVENTIONS:
Diagnostic Test: collection of expectoration, stools and blood — collection of expectoration, stools and blood

SUMMARY:
The objective of this study is to evaluate the predictive nature of the biomarker Porphyromonas catoniae measured at the age of 12 months in the occurrence of colonization with Pseudomonas aeruginosa at 36 months of age in children with cystic fibrosis.

DETAILED DESCRIPTION:
This is a multicentric study in 3 phases:

* Pre-inclusion: at the first visit to the CRCM (support for a positive screening confirmed by sweat test and genotyping CFTR)
* Inclusion: possible between the 2nd visit to the CRCM (about 2 months old) and the 6th month
* Follow-up: up to 36 months old. The pace of visits will be based on the usual follow-up rate of CF infants

The clinical data as well as samples (expectorations, stools) will be collected on a monthly basis up to 6 months old and then every 2 months until one year old and finally quarterly until 3 years old.

* Tracheo-bronchial secretions will be collected at the CRCM
* Stools samples will be carried out by the parents prior to consultation with the CRCM
* A blood collection will be carried out annually in an annual report.

ELIGIBILITY:
Inclusion criteria:

* Infants aged 6 months maximum at inclusion with a confirmed diagnosis of cystic fibrosis in its classical form (positive sweat test and/or two mutations of the CFTR gene from class I to III)
* Children free from any antecedent of colonization to P. aeruginosa at the time of inclusion (certified by the microbiological history supplemented by a molecular test by qPCR according to the diagram of Le gal et al., 2013)-Affiliation to the social security system
* Consent signed by the holders of parental authority or the sole parent holding parental authority / and "oral" agreement of the second holder

Exclusion criteria:

* Severe acute pathology (other than cystic fibrosis) in progress, or requiring surgery
* Children unable to undergo the tests required for the Protocol
* Children whose parent (s) is (are) minor (s)
* Children whose parental authority does not master the French language
* Refusal to participate in the study

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Presence of P. aeruginosa in bacterial sputum cultures collected at 36 months of age | 36 months
  positive or negative

SECONDARY OUTCOMES:
Absolute amount of P. aeruginosa at different sampling times. | 36 months
  amount (UFC/mL)
Absolute amount of P. catoniae in respiratory secretions at different sampling times and Delta between 12, 24 and 36 months. | 36 months
  amount (UFC/mL)
Absolute amount of P. catoniae in stool at different sampling times and Delta between 12, 24 and 36 months. | 36 months
  amount (UFC/mL)
Level of dysbiosis | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve HERY-ARNAUD, Pr, Principal Investigator — University Hospital, Brest
Locations (11):
- France (11):
  - CHRU Angers, Angers
  - Hôpital des Enfants Bordeaux, Bordeaux
  - CHU Grenoble, Grenoble
  - Hôpital Femme-Mère-Enfant Lyon, Lyon
  - CHRU Nantes, Nantes
  - Hôpital Necker, Paris
  - Hôpital Trousseau, Paris
  - CHRU Rennes, Rennes
  - Centre de Perharidy, Roscoff
  - Hôpital Charles Nicolle Rouen, Rouen
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.